CLINICAL TRIAL: NCT06431399
Title: A Randomized, Open-label, Crossover Phase 1 Clinical Trial to Evaluate the Safety, Pharmacokinetic Characteristics and the Effect of Food After Administration of JLP-2004 in Healthy Adult Volunteers
Brief Title: To Evaluate the Safety, Pharmacokinetic Characteristics and the Effect of Food After Administration of JLP-2004
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JP-2004-102
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JLP-2004 FAST (Experimental): Thin arm is JLP-2004 FAST condition
  Interventions: Drug: JLP-2004 qd
- JLP-2004 FED (Experimental): Thin arm is JLP-2004 FED condition
  Interventions: Drug: JLP-2004 qd

INTERVENTIONS:
Drug: JLP-2004 qd — Group I(Peroid I-JLP-2004 FAST, Peroid II-JLP-2004 FED), Group II(Period I-JLP-2004 FED, Period II-JLP-2004 FAST)
  Other Names: painkiller

SUMMARY:
To evaluate the safety, pharmacokinetic characteristics and the effect of food after administration of JLP-2004

DETAILED DESCRIPTION:
A randomized, open-label, crossover phase 1 clinical trial to evaluate the safety, pharmacokinetic characteristics and the effect of food after administration of JLP-2004 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 years or older at the time of screening
2. At the time of screening, those who weigh more than 50.0 kg and have a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less.
3. Those who do not have congenital or chronic diseases and have no pathological symptoms or findings as a result of internal medical examination (if necessary, electroencephalography, electrocardiogram, chest and stomach endoscopy, or gastrointestinal radiography)
4. Those who be considered suitable for clinical subjects according to the results of laboratory tests (hematology tests, blood chemistry tests, urine tests, serum tests, blood coagulation tests, urine drugs tests), physical examinations and 12-lead electrocardiography at the time of screening
5. Those who voluntarily decide to participate and agree in writing to comply with the subject compliance requirements during the clinical trial period after receiving a detailed explanation of this clinical trial and fully understanding it

Exclusion Criteria:

1. Those who have current or past medical history of clinically significant liver, kidney, nervous system, mental, respiratory, endocrine, blood disease, tumor, genitourinary, cardiovascular, digestive, and musculoskeletal systems, as well as the following symptoms or history.

   ① Renal impairment

   ② Liver disorder
2. For women, pregnant women (Urine-HCG positive) or breastfeeding mother
3. Those who have clinically significant hypersensitivity reactions such as asthma, hives, allergies, etc. to the main ingredient (Pelubiprofen), additives, or other drugs (aspirin or other non-steroidal anti-inflammatory drugs (including COX-2 inhibitors)) and have a history of hypersensitivity reaction
4. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
5. Those with a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of clinical trial drugs

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
AUCt of JLP-2004 | after treatment 0hour, 0.5hour, 1hour, 2hour, 3hour, 24hour
  AUCt of JLP-2004 in FAST and FED condition
Cmax of JLP-2004 | after treatment 0hour, 0.5hour, 1hour, 2hour, 3hour, 24hour
  Cmax of JLP-2004 in FAST and FED condition

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Park, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Chungju, Seowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No